CLINICAL TRIAL: NCT01409343
Title: A Phase I Dose-Escalation and Pharmacokinetic Study of TrasGEX™ in Patients With Locally Advanced or Metastatic HER-2-positive Cancer
Brief Title: TrasGEX™: Phase 1 Study in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glycotope GmbH (Industry)
Collaborators: Glycotope Biotechnology GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEXMab73101
Record Dates: First submitted 2011-07-18; First posted 2011-08-04 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Solid Tumors
Keywords: advanced solid cancers; metastatic solid cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TrasGEX (Experimental): A total of 37 patients with advanced HER2-positive carcinomas and progressive disease.
  Interventions: Drug: TrasGEX™

INTERVENTIONS:
Drug: TrasGEX™ — Patients received TrasGEX intravenously every 3 weeks until disease progression in doses of 12-720 mg in a three-plus-three dose escalation design, including an expansion cohort at the highest dose.

SUMMARY:
This was a prospective, open label, multicenter study evaluating the safety, tolerability and pharmacokinetics of TrasGEX™ after intravenous administration in patients with HER-2 positive cancers. The effect of TrasGEX™ on the development of anti-drug antibodies and on tumour response was also evaluated.

DETAILED DESCRIPTION:
Adult patients with advanced and/or metastatic HER2-positive cancer who were resistant to or for whom there was no standard anti-tumor therapy available at the time of enrollment and who had an estimated life expectancy of at least 3 months were eligible for participation in this study.

Patients were to receive the study drug until disease progression (clinical or radiologic), unacceptable toxicity, or any other reason leading to termination of study treatment.

Dose-escalation was performed in 3 to 6-patient cohorts.

ELIGIBILITY:
Main Inclusion Criteria:

1. Signed written informed consent granted prior to initiation of any study-specific procedures;
2. Male or female patients of ≥18 years of age;
3. ERBB2 (HER-2) gene amplification or ERBB2 overexpression
4. Histologically or cytologically confirmed cancer, either locally advanced or metastatic;
5. No anti-tumor therapy of proven benefit available at study enrollment;
6. Life expectancy of >=3 months;
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) <=2;
8. Male or female patients of child-producing potential must agree to use contraceptive measures or oral contraception during the study and for 28 days after the last dose of TrasGEX™;
9. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of TrasGEX™;

and

Main Exclusion Criteria:

1. Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within 4 weeks of the first dose of TrasGEX™;
2. Major surgery within four weeks of the first dose of TrasGEX™;
3. Newly diagnosed brain metastases, metastases that have been documented to be stable for <3 months, or metastases for which systemic corticosteroids are required;
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition as TrasGEX™;
5. History of myocardial infarction within 12 months of the administration of the first dose of TrasGEX™;
6. History of congestive heart failure defined as Class II to IV per New York Heart Association classification within 12 months of the administration of the first dose of TrasGEX™;
7. Left ventricular ejection fraction <50%;
8. Previous malignancy other than the current diagnosis within 5 years of the first dose of TrasGEX™;
9. Pregnancy or lactation; and
10. Concurrent uncontrolled significant illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
optimal dose and regimen of TrasGEX™ | up to at least 8 weeks after the first TrasGEX™ administration
  The primary objective of this first-in-man study is to determine the optimal dose and regimen of TrasGEX™ in patients with locally advanced or metastatic human epidermal growth factor receptor-2 (HER-2)-positive cancer. The recommended phase II dose needs to have an acceptable safety profile and provides evidence for efficacy based on clinical observations or the pharmacokinetic profile.

SECONDARY OUTCOMES:
To determine preliminary evidence of activity | approx. every 8 weeks
  CT or MRI imaging will be performed. Assessment of tumor response (SD, PR, CR. PD) will be performed following a modified version of the revised RECIST guidelines, version 1.1. Basically, patients will receive treatment with TrasGEX™ until progression of disease and/or unacceptable toxicities are observed.
safety and tolerability of TrasGEX™ | until 4 weeks after the last treatment with TrasGEX™
  To assess the safety and tolerability of TrasGEX™ in patients with advanced and/or metastatic HER-2-positive cancer at various dose levels considering observed adverse events, laboratory values, vital signs, ECOG performance status and physical examination.
To assess the pharmacokinetic (PK) profile of TrasGEX™ (part I) | prior to 1st infusion until the end of 5th infusion
  c(max): to determine the PK profile samples will be taken before the first infusion and up to 24 h after after infusion, followed by weekly samples for the first infusion and samples immediately before and after infusion for the following infusions
To assess the pharmacokinetic (PK) profile of TrasGEX™ (part II) | prior to 1st infusion until the end of 5th infusion
  t(1/2): to determine the PK profile samples will be taken before the first infusion and up to 24 h after after infusion, followed by weekly samples for the first infusion and samples immediately before and after infusion for the following infusions

CONTACTS AND LOCATIONS:
Overall Officials: Glycotope GmbH, Study Director — Glycotope GmbH
Locations (5):
- Austria (2):
  - Glycotope Investigational Site, Graz
  - Glycotope Investigational Site, Innsbruck
- Glycotope Investigational Site, Hamburg, Germany
- Glycotope Investigational Site, Milan, Italy
- Glycotope Investigational Site, Bellinzona, Switzerland

REFERENCES:
- [Result] Fiedler W, Stoeger H, Perotti A, Gastl G, Weidmann J, Dietrich B, Baumeister H, Danielczyk A, Goletz S, Salzberg M, De Dosso S. Phase I study of TrasGEX, a glyco-optimised anti-HER2 monoclonal antibody, in patients with HER2-positive solid tumours. ESMO Open. 2018 Jun 23;3(4):e000381. doi: 10.1136/esmoopen-2018-000381. eCollection 2018. PMID 30018811